CLINICAL TRIAL: NCT03361696
Title: Development, Optimization, Efficiency of the Interface System of Communication and Control of the Environment
Acronym: DOME-6
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-112
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2017-11

CONDITIONS: Handicaps Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Help to use the Interface System of Communication and Control of the Environment — the occupational therapist and the ergonomics engineers at the rate of 4 sessions per patient for periods of 2 to 3 hours help patient to use use the Interface System of Communication and Control of the Environment

SUMMARY:
The objective of this project is the realization of tests at home and in Hospitals or Functional Rehabilitation for the improvement of the communication with the family and medical entourage, the facility of the emotional expression, the evaluation of the pain, the control of home automation to increase their autonomy, facilitated their reintegration at home. The work is the last step of the research program started in 2009, with the optimization of the installation of the system, the improvement of physical and computer ergonomic aspects and the development of dedicated interfaces according to the type of disability and needs. of each one.

A work upstream of the definition of specifications taking into account the medical constraints was realized and the actions of improvement of the models, the algorithms, the robustness and the effectiveness of the treatment are in progress . The specific adaptation to concrete cases should lead to a system that allows 90% of the population of people with disabilities to exploit the system and significantly improve their level of communication, autonomy and in fact their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Patients (2-80 years old) with complete or near complete motor disability of both upper limbs or four limbs: Sequelae of trauma or advanced rheumatologic disease (spinal cord injury, upper limb amputation, head trauma, chronic polyarthritis), Diseases Congenital (myopathies, agenesis upper limbs), sequelae of vascular accident (medullary infarction, syringomyelia), neurodegenerative diseases (amyotrophic lateral sclerosis, multiple sclerosis, conduction block neuropathy, etc ..).
* Patients older than 55 years without disability but with a loss of dependence.
* Troubles of the communication and loss of autonomy.

Exclusion Criteria:

* Patient with severe visual contraindications (decreased visual acuity with correction of ± 6/7 dioptres, major oculomotor abnormalities).
* Patients with significant cognitive impairment to understand simple instructions related to the use of the system

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe disabilities either of traumatic origin or of neurological origin or Patients over 55 with loss of autonomy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Quality of life questionnaire SF36 | change over baseline and end of follow-up at 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No